CLINICAL TRIAL: NCT02913638
Title: A Post-Breastfeeding Intervention Observational Follow-Up Study
Brief Title: A Post Breastfeeding Follow-Up Study
Status: Completed | Type: Observational
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Sponsor
Other Study IDs: AL08X
Record Dates: First submitted 2016-09-07; First posted 2016-09-26 (Estimated); Last update posted 2017-02-13 (Actual); Status verified 2017-02

CONDITIONS: Breast Feeding
MeSH Terms: conditions — Breast Feeding

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this clinical study which is to evaluate the benefits of lactation support intervention, in conjunction with maternal nutritional supplementation during the last trimester to 12 weeks postpartum in comparison to pre- and postnatal care on 1) breast feeding practices (primary objective), and 2) cognitive development in children within 28 months 16 days - 32 months 30 days (secondary objective).

DETAILED DESCRIPTION:
This is an observational study involving mothers and their child at 30 months old as a follow up to the breastfeeding intervention study that they have participated in and completed during the period from the last trimester to 12 weeks postpartum.

The assessors will be blinded to subject's treatment group assignment from the intervention phase.

There are no products given to any subject.

The primary variable is duration of any breastfeeding from birth.

ELIGIBILITY:
Inclusion Criteria:

* Mother and child pair was enrolled in and completed the breastfeeding intervention (AL08) study.
* Age of child is within the allowable window (28 months 16 days - 32 months 30 days).
* Subject's parent/Legally Acceptable Representative (LAR) is willing and able to follow study procedures.
* Subject's parent/LAR has voluntarily signed and dated an Informed Consent Form (ICF), approved by an Independent Ethics Committee/Institutional Review Board (IEC/IRB) or other applicable privacy regulation authorization prior to any participation in the study.

Exclusion Criteria:

* Child has a diagnosis of developmental disorders e.g. cerebral palsy that require medical intervention prior to enrollment in this study.

Ages: 28 Months to 32 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study involves mothers and their child at 30 months old as a follow up to the breastfeeding intervention study that they have participated in and completed during the period from the last trimester to 12 weeks postpartum
Sampling Method: Probability Sample
Enrollment: 196 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Duration of any breastfeeding from birth | 32 months
  The primary variable, which is the duration of any breastfeeding from birth, will be assessed in all mothers recruited for this study. A questionnaire will be used to capture information on the age of the child (in months/weeks) in which the mother stopped breastfeeding. This information will be used to derive any breastfeeding duration from birth onwards.

SECONDARY OUTCOMES:
Cognitive outcomes | 32 months
  Bayley Scales (BSID-III) of Infant and Toddler Development
Language/Communication outcomes | 32 months
  Age & Stages Questionnaire (ASQ-3)

CONTACTS AND LOCATIONS:
Overall Officials: Dieu Huynh, M.D., Study Chair — Abbott Nutrition
Locations (4):
- Vietnam (4):
  - An Lao District Health Center, Haiphong
  - Binh Luc District Health Center, Hà Nam
  - Yen Mo District Health Center, Ninh Bình
  - Phu Binh District Health Center, Thái Nguyên

IPD SHARING:
Plan to Share IPD: No